CLINICAL TRIAL: NCT04308291
Title: The MiniMed™ 780G Glycemic Control and Quality of Life Study for the Treatment of Pediatric and Adult Subjects With Type 1 Diabetes in France (EQOL Study)
Brief Title: The MiniMed™ 780G Glycemic Control and Quality of Life Study for the Treatment of Pediatric and Adult Subjects With Type 1 Diabetes in France.
Status: Completed | Type: Observational
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP328
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-01

CONDITIONS: Type 1 Diabetes
Keywords: 780G, T1D
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- MiniMed™ 780G System: Subject will use the MiniMed™ 780G System as per standard of care.
  Interventions: Device: MiniMed™ 780G System

INTERVENTIONS:
Device: MiniMed™ 780G System — Subject enrolled in the study will start using the MiniMed™ 780G pump in Auto Mode after a run-in period of two weeks in Manual Mode (with no SmartGuard™ functions). Study phase in Automode will follow a 6 and 12 months follow- up as per standard of care.

SUMMARY:
The purpose of the study is to evaluate the efficacy in glycemic control and the impact on the quality of life of patients using the MiniMed™ 780G System for the treatment of Type 1 diabetes, in real life settings in France.

DETAILED DESCRIPTION:
Local, post-market, non-interventional, prospective, single-arm, multi-center study of patients pediatric and adult.

The study is conducted according to the same schedule as the routine follow-up of patients:

1. RUN-IN PHASE: Subject will start a run-in phase in an out of hospital setting, as per standard practice of the site. The objective of the run-in phase is to train the subjects on the MiniMed™ 780G insulin pump, assess subjects' compliance and ability to comprehend the study procedures and tolerance of wearing the sensor and transmitter continuously. It is expected that during the run-in phase the MiniMed™ 780G insulin pump will be set in Manual mode and all the algorithms are switched off, and baseline Continuous Glucose Monitoring (CGM) data will be collected. The expected duration of the run-in phase is approximately 2 weeks. At the end of the run-in phase the MiniMed™ 780G insulin pump will be set in Auto Mode and the date of activation will be collected and identified as a start of the study phase. Data from the MiniMed™ 780G insulin pump will be uploaded in the CareLink™ as per standard practice, before Auto Mode activation.
2. 6 AND 12 MONTHS FOLLOW UP: Follow-up visits will be performed according to the therapy management standard of care at 6 and 12 months after Auto Mode activation in the study.

Approximately 300 patients (children and adults) will be enrollment in the study in approximately 32 sites in France.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥7 years of age.
2. Subject has a clinical diagnosis of type 1 diabetes for more than 1 year as determined via medical records or source documentation by an individual qualified to make a medical diagnosis.
3. Subject has a HbA1c value greater than 6.5% and less than 12% at time of enrolment visit.
4. Subject is under Continuous Subcutaneous Insulin Infusion (CSII) therapy (with or without Continuous Glucose Monitoring) ≥ 6 months before enrolment.
5. Subject requires ≥8 units of insulin per day.
6. Subjects and their parent(s)/guardian(s) must be able to speak and be literate in French as verified by the investigator.
7. Subjects and their parent(s)/guardian(s) are willing to participate in the study and sign the Data Release Form (DRF).
8. Subjects who are ≥18 years of age should be able to provide consent.

Exclusion Criteria:

1. Subject has MiniMed™ 780G System IFU contraindication(s).
2. Subject uses Predictive Low-Glucose Management (PLGM) System (i.e. MiniMed™ 640G with SmartGuard) in the last 6 months before the enrolment.
3. Subject uses Low Glucose suspend (LGS) feature (i.e. MiniMed™ Paradigm Veo Pump) in the last 6 months before the enrolment.
4. Subject under Multiple-Daily Injections (MDI) treatment in the 6 months before the enrolment.
5. Subject has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).

Min Age: 7 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects 7 years of age or older with T1D and under Continuous Subcutaneous Insulin Infusion (CSII) therapy (with or without CGM)
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- France (32):
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - APHP Avicenne, Bobigny
  - CHU Bordeaux (Saint-André), Bordeaux
  - CH Boulogne-Sur-Mer, Boulogne-sur-Mer
  - CHU Brest, Brest
  - HCL Groupement Hospitalier Est, Bron
  - CHU Caen, Caen
  - Ch Sud Francilien, Corbeil-Essonnes
  - CHU Dijon, Dijon
  - CHRU La Rochelle, La Rochelle
  - CHU Grenoble, La Tronche
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - HCL DIAB-eCARE, Lyon
  - IDNC Chartres, Mainvilliers
  - APHM Marseille (Hôpital de la Conception), Marseille
  - APHM Marseille (La Timone), Marseille
  - GHEF (Centre Hospitalier de Meaux), Meaux
  - CHU Montpellier (Lapeyronie), Montpellier
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU Nîmes, Nîmes
  - APHP Bichat, Paris
  - APHP Cochin, Paris
  - Ch Lariboisiere, Paris
  - CH Perpignan, Perpignan
  - CH Périgueux, Périgueux
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse (Rangueil), Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kessler L, Thivolet C, Penfornis A, Gouet D, Coffin C, Moret M, Borot S, Bekka S, Sonnet E, Joubert M, Lablanche S, Burtin G, Di Piazza F, van den Heuvel T, Cohen O. Advanced Hybrid Closed Loop Algorithm Use in Type 1 Diabetes: The French MiniMed Glycemic Control and Quality of Life Study. Diabetes Ther. 2025 Mar;16(3):413-427. doi: 10.1007/s13300-024-01673-9. Epub 2024 Dec 17. PMID 39688775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first subject enrollment: 15-FEB-2021, Date of last data received: 23-NOV-2022
Pre-assignment Details: 306 subjects with type 1 diabetes consented to participate in the study. Of them, 16 subjects are Screen Failure.
Period: Run-In Phase
Arm/Group | MiniMed™ 780G System
Started | 290
Completed | 286
Not Completed | 4
Not completed — Withdrawal by Subject | 4
Period: Study Phase 6-M
Arm/Group | MiniMed™ 780G System
Started | 286
Completed | 270
Not Completed | 16
Not completed — Withdrawal by Subject | 13
Not completed — Physician Decision | 2
Not completed — Carelink uploading issues (Linux user) | 1
Period: Study Phase 12-M
Arm/Group | MiniMed™ 780G System
Started | 270
Completed | 256
Not Completed | 14
Not completed — Withdrawal by Subject | 11
Not completed — Physician Decision | 2
Not completed — Hospitalization for cause not related to the study (Pancytopenia) | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects, excluding Screen Failure
Arm/Group | MiniMed™ 780G System
Number analyzed (Participants) | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (16.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160
  Male | 130
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 290
HbA1c [Mean (Standard Deviation); unit: %] — Population: 2 subjects, out of 290, with missing HbA1c information at baseline
  %
    number analyzed (Participants) | 288
    (all) | 7.76 (0.818)

OUTCOME MEASURES:

1. Primary Outcome: Time in Range 70-180 mg/dL (TIR)
Description: The change in (%) the time spent within range, defined as the proportion of sensor glucose concentration within the target range of 70-180 mg/dL, between baseline and 6 months.
Time Frame: 0-6 months
Population: Out of 290 subjects enrolled (excluding screen failure), 263 subjects, with both baseline and 6-M Follow Up measurements available were included in the analysis
Measure: Mean (95% Confidence Interval); unit: % of time
Arm/Group | MiniMed™ 780G System
Number analyzed (Participants) | 263
% of time | 11.81 [10.72 to 12.90]
Statistical Analysis 1: Comparison: MiniMed™ 780G System; Test type: Superiority; p < 0.0001, t-test, 2 sided; paired t-test

2. Secondary Outcome: Satisfaction Score
Description: To evaluate the change from baseline in satisfaction score based on the Diabetes Treatment Satisfaction Questionnaire change (DTSQc)
Time Frame: 0-6 months
Reporting Status: Not Posted

3. Secondary Outcome: Quality of Life Change
Description: To evaluate the change in quality of life based on the Diabetes Quality of life questionnaire (DQoL)
Time Frame: 0-6 months
Reporting Status: Not Posted

4. Secondary Outcome: Fear of Hypoglycemic Events Change
Description: To evaluate the change from baseline in the fear of hypoglycemic events based on the Hypoglycemia Fear Survey (HFS)
Time Frame: 0-6 months
Reporting Status: Not Posted

5. Secondary Outcome: Treatment Satisfaction Score
Description: To evaluate the treatment satisfaction score based on the Diabetes Treatment Satisfaction Questionnaire status (DTSQs)
Time Frame: 0-6 months
Reporting Status: Not Posted

6. Secondary Outcome: Glycemic Parameters Changes
Description: To evaluate the change in glycemic parameters: mean time of sensor glucose values below 70mg/dL
Time Frame: 0-6 months
Reporting Status: Not Posted

7. Secondary Outcome: Glycemic Parameters Changes
Description: To evaluate the change in glycemic parameters: mean time of sensor glucose values below 54mg/dL
Time Frame: 0-6 months
Reporting Status: Not Posted

8. Secondary Outcome: Glycemic Parameters Changes
Description: To evaluate the change in glycemic parameters: mean time of sensor glucose values above 180mg/dL
Time Frame: 0-6 months
Reporting Status: Not Posted

9. Secondary Outcome: Glycemic Parameters Changes
Description: To evaluate the change in glycemic parameters: mean time of sensor glucose values above above 250mg/dL
Time Frame: 0-6 months
Reporting Status: Not Posted

10. Secondary Outcome: HbA1c
Description: To evaluate the change in glycosylated haemoglobin (HbA1c), between baseline and 6 months.
Time Frame: 0-6 months
Measure: Mean (Standard Deviation); unit: Hba1c %
Arm/Group | MiniMed™ 780G System
Number analyzed (Participants) | 264
Hba1c % | -0.52 (0.719)

11. Secondary Outcome: Time in Range of 70-180 mg/dL (TIR)
Description: The change in (%) the time spent within range, defined as the proportion of sensor glucose concentration within the target range of 70-180 mg/dL, between baseline and 12 months.
Time Frame: 0-12 months
Measure: Mean (95% Confidence Interval); unit: % of time
Arm/Group | MiniMed™ 780G System
Number analyzed (Participants) | 256
% of time | 11.09 [10.37 to 11.82]

12. Secondary Outcome: HbA1c
Description: To evaluate the change in glycosylated haemoglobin (HbA1c), between baseline and 12 months.
Time Frame: 0-12 months
Measure: Mean (Standard Deviation); unit: Hba1c %
Arm/Group | MiniMed™ 780G System
Number analyzed (Participants) | 251
Hba1c % | -0.42 (0.754)

ADVERSE EVENTS:
Description: Adverse Events were not collected. For this reason we reported 0/0 in the mandatory numeric fields below.
Arm/Group | MiniMed™ 780G System
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT04308291/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT04308291/SAP_001.pdf